CLINICAL TRIAL: NCT03329417
Title: Effects of a Virtual Reality-Based Mirror NeuroRehabilitation System (VR-based MNRS) on Functional Performance of Upper Extremity for Unilateral Stroke Patients
Brief Title: Neurorehabilitation Using a Virtual Reality-based Mirror Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-105-213
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-03

CONDITIONS: Rehabilitation, Mirror Neurons, Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional occupational therapy (Active Comparator): The program includes 30 minutes of traditional occupational therapy (sensorimotor facilitation techniques, such as: Rood, Bobath and propriocetive-neuromuscular-facilitation), followed by 20 minutes of motor task specific training in each treatment session.
  Interventions: Other: task-oriented training
- Mirror therapy using a mirror box (Active Comparator): The program includes 30 minutes of mirror therapy, followed by 20 minutes of regular motor task specific training in each treatment session.
  Interventions: Other: task-oriented training
- Virtual reality based mirror therapy (Experimental): The program includes 30 minutes treatment session of virtual reality mirror therapy, followed by 20 minutes of motor task specific training in each treatment session.
  Interventions: Other: task-oriented training

INTERVENTIONS:
Other: task-oriented training — Motor training targeted to goals that are relevant to the functional needs of the patient

SUMMARY:
In the proposed study, the investigators assumed that mirror therapy combined with virtual reality technology will provide a better treatment effects than traditional mirror therapy for the patients with unilateral stroke. The aim of the study is to examine the difference in the treatment effects among the combination of task-oriented training with either virtual reality based mirror therapy, mirror therapy or traditional occupational therapy on the upper extremity function and brain activity of the stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of stroke with unilateral side involved;
2. A score of Mini-mental state examination greater than 24 for proving higher mental function;
3. Time of onset > 6 months before treatment begins, and
4. Premorbid right-handedness.

Exclusion Criteria:

1. Vision loss;
2. Major cognitive-perceptual deficit;
3. Other brain disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Change in the result of Fugl-Meyer assessment (FMA) for motor function of upper extremity test | baseline, 6 weeks and 18 weeks
  Each item is rated on a three-point ordinal scale (2 points for the detail being performed completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.
Change in the result of Modified Ashworth scale (MAS) | baseline, 6 weeks and 18 weeks
  Muscle tone is defined by the resistance of a muscle being stretched without resistance. The MAS scores were distributed across the entire scale, ranging from 0 to 4, that is convenient for the clinician use. The grading of the scale is described as below: 0) no increase in muscle tone; 1) minimal resistance at the end of the range of motion; 1+) slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the reminder (less than half) of the ROM; 2) more marked increase in tone but only after part is easily flexed; 3) considerable increase in tone; and 4) passive movement is difficult and affected part is rigid in flexion or extension.
Change in the result of Box and blocks test | baseline, 6 weeks and 18 weeks
  The score is the number of blocks carried from one box to the other in one minute. Higher values represent a better outcome.
Change in the result of Semmes-Weinstein monofilament (SWM) test | baseline, 6 weeks and 18 weeks
  The Semmes-Weinstein monofilamenttest examines the cutaneous pressure threshold, range from 1.65-6.65. Higher values represent a worse outcome.
Change in the result of Motor Activity Log | baseline, 6 weeks and 18 weeks
  Semi-structured interview examine how much and how well the subject uses their more-affected arm for 30 ADLs. Score range from 0-180. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Change in Power Spectrum of the Electroencephalography (EEG) | baseline and 6 weeks
  Power spectrum is computed for the alpha (8-13 Hz) and beta (14-24 Hz) frequency bands. Higher values represent a better outcome.
Changes in Cortical Excitability Assessed by Transcranial Magnetic Stimulation | baseline and 6 weeks
  Cortical silent period of to evaluate intercortical facilitation of brain. Lower values represent a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Hsu HY, Kuo LC, Lin YC, Su FC, Yang TH, Lin CW. Effects of a Virtual Reality-Based Mirror Therapy Program on Improving Sensorimotor Function of Hands in Chronic Stroke Patients: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2022 Jun;36(6):335-345. doi: 10.1177/15459683221081430. Epub 2022 Mar 28. PMID 35341360